CLINICAL TRIAL: NCT04726917
Title: Assessment of Stress Levels and Depressive and Anxiety Symptoms in Patients With COPD During In-Hospital Pulmonary Rehabilitation: An Observational Cohort Study
Brief Title: Assessment of Stress Levels and Depressive and Anxiety Symptoms in Patients With COPD
Status: Completed | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: OpoleUofTech4
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: COPD; Anxiety State; Stress; Depressive Symptoms; Mood Disorders
Keywords: pulmonary rehabilitation; depression; anxiety; stress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COPD: Patients qualified for 3-week in-hospital pulmonary rehabilitation
  Interventions: Behavioral: Pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — Patients qualified for rehabilitation were assessed for stress levels as well as symptoms of anxiety and depression before rehabilitation began

SUMMARY:
The aim of the study was to assess the levels of depression, anxiety and stress in patients with COPD qualified for In-hospital pulmonary rehabilitation program

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), manifested by coughing, shortness of breath, sputum production, wheezing and reduced physical performance, is one of the most frequently diagnosed lung diseases. Anxiety and depression have been found to increase the number of acute exacerbations and hospitalizations (thus reducing quality of life), weight, appetite, sleep disorders, fatigue or loss of energy, lack of concentration, pessimism about the future and suicidality. Anxiety has been estimated to occur in 21-96% and depression in 27-79% of patients with COPD, values that are higher than for the general population or other chronic diseases. Pulmonary rehabilitation leads to the improvement to the physical capacity and overall fitness of the patients with COPD allowing restoration of independence in daily functioning. Psychological support is required in order to reduce the negative psychological symptoms related to both the pulmonary disease itself and the comorbidities. In the presented study, the aim was to assess the prevalence of levels of depression, anxiety and stress in patients with COPD qualified for In-hospital pulmonary rehabilitation program.

The program includes the following elements:

Three weeks of pulmonary rehabilitation conducted in an outpatient care facility:

* 5- time a week for 30 minutes a specific respiratory exercises- relaxation exercises for breathing muscles, exercises to increase breathing, prolonged exhalation exercise, chest percussion
* 5- time a week for 20-30 min training on a cycle ergometer
* 5- time a week for 30 minutes a fitness and respiratory exercises - coordination and balance exercises, stretching exercises
* relaxation training by Schultz. The technique involves the daily practice of sessions that last around 15 minutes. During each session, the practitioner repeats a set of visualisations that induce a state of relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as COPD;
* Pulmonary rehabilitation conducted in ward settings;

Exclusion Criteria:

* inability to self-complete the research questionnaires;
* presence of the following issues at the time of the examination or in the medical data: disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders;
* initiation of psychiatric treatment during the research project;
* the patient's refusal at any stage of the research project.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.
Perception of Stress Questionnaire (PSQ) | 30 minutes
  The Perception of Stress Questionnaire (PSQ) is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | 10 minutes
  The six-minute walk test measures the distance a patient is able to walk over a total of six minutes on a firm, flat surface. The aim is for the patient to walk as far as possible in six minutes. The patient is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Spirometry Test | 20 minutes
  The patient is asked to take the deepest breath they can, and then exhale into the sensor as hard as possible, for as long as possible, preferably at least 6 seconds. It is sometimes directly followed by a rapid inhalation, in particular when assessing possible upper airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Szczegielniak, Prof, Study Chair — Hospital of Ministry of the Interior and Administration
Locations (1):
- Hospital of Ministry of the Interior and Administration, Głuchołazy, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tselebis A, Bratis D, Pachi A, Moussas G, Ilias I, Harikiopoulou M, Theodorakopoulou E, Dumitru S, Kosmas E, Vgontzas A, Siafakas N, Tzanakis N. A pulmonary rehabilitation program reduces levels of anxiety and depression in COPD patients. Multidiscip Respir Med. 2013 Jun 22;8(1):41. doi: 10.1186/2049-6958-8-41. PMID 23931626
- [Background] Bhandari NJ, Jain T, Marolda C, ZuWallack RL. Comprehensive pulmonary rehabilitation results in clinically meaningful improvements in anxiety and depression in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil Prev. 2013 Mar-Apr;33(2):123-7. doi: 10.1097/HCR.0b013e31828254d4. PMID 23399845
- [Background] da Costa CC, de Azeredo Lermen C, Colombo C, Canterle DB, Machado ML, Kessler A, Teixeira PJ. Effect of a Pulmonary Rehabilitation Program on the levels of anxiety and depression and on the quality of life of patients with chronic obstructive pulmonary disease. Rev Port Pneumol. 2014 Nov-Dec;20(6):299-304. doi: 10.1016/j.rppneu.2014.03.007. Epub 2014 May 27. PMID 24874610
- [Background] Luk EK, Gorelik A, Irving L, Khan F. Effectiveness of cognitive behavioural therapy in a community-based pulmonary rehabilitation programme: A controlled clinical trial. J Rehabil Med. 2017 Mar 6;49(3):264-269. doi: 10.2340/16501977-2189. PMID 28150856
- [Background] Coventry PA, Bower P, Keyworth C, Kenning C, Knopp J, Garrett C, Hind D, Malpass A, Dickens C. The effect of complex interventions on depression and anxiety in chronic obstructive pulmonary disease: systematic review and meta-analysis. PLoS One. 2013 Apr 5;8(4):e60532. doi: 10.1371/journal.pone.0060532. Print 2013. PMID 23585837
- [Background] Zhang MW, Ho RC, Cheung MW, Fu E, Mak A. Prevalence of depressive symptoms in patients with chronic obstructive pulmonary disease: a systematic review, meta-analysis and meta-regression. Gen Hosp Psychiatry. 2011 May-Jun;33(3):217-23. doi: 10.1016/j.genhosppsych.2011.03.009. Epub 2011 Apr 27. PMID 21601717
- [Background] Panagioti M, Scott C, Blakemore A, Coventry PA. Overview of the prevalence, impact, and management of depression and anxiety in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Nov 13;9:1289-306. doi: 10.2147/COPD.S72073. eCollection 2014. PMID 25419126